CLINICAL TRIAL: NCT04142333
Title: GIA in Cascade Testing
Acronym: GIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Kari Ring, MD, Assistant Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 21168
Record Dates: First submitted 2019-07-18; First posted 2019-10-29 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Genetic Predisposition
Keywords: genetic counseling; genetic testing
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GIA Access (Other): All patients consented to this study will be given access to the GIA technology to share with their family members.
  Interventions: Genetic: GIA

INTERVENTIONS:
Genetic: GIA — Patients receive a secure GIA link from their provider and then are able to send their relatives the link to GIA through texting, email, and/or Facebook messenger. Once a relative clicks on the provided link, GIA's platform is structured as a decision tree, allowing family members to construct a personalized conversation about their family member's test results. This can be done either on a smartphone or computer. GIA provides basic genetics education and risk assessment and connects family members with local genetic counseling resources to continue this conversation and/or go forward with genetic testing. At the end of the conversation, the family member has the option of having a transcript sent to them via email for their reference. The objective of the current study is to evaluate the application of GIA for cascade testing in newly identified high risk breast and gynecologic mutation carriers.

SUMMARY:
The objective of this pilot study is to evaluate the feasibility and acceptability of GIA in sharing genetic test results with family members.

To determine the utility of GIA in sharing information. To determine the impact of GIA on downstream cascade testing rates.

DETAILED DESCRIPTION:
Chatbots, also known as conversation agents, are programs designed to have interactive conversations with humans. While traditionally used in sectors such as online gaming and customer service, chatbots have made their way into a number of industries including healthcare and have shown promise in areas such as managing anxiety/depression, weight loss, and medication adherence. GIA (Genetic Information Assistant) is a chatbot specifically designed as a tool for patients to use for disseminating genetic results, education, and genetic counseling resources to their family members after they themselves receive a positive result.

Patients receive a secure GIA link from their provider and then are able to send their relatives the link to GIA through texting, email, and/or Facebook messenger. Once a relative clicks on the provided link, GIA's platform is structured as a decision tree, allowing family members to construct a personalized conversation about their family member's test results. This can be done either on a smartphone or computer. GIA provides basic genetics education and risk assessment and connects family members with local genetic counseling resources to continue this conversation and/or go forward with genetic testing. At the end of the conversation, the family member has the option of having a transcript sent to them via email for their reference. The objective of the current study is to evaluate the application of GIA for cascade testing in newly identified high risk breast and gynecologic mutation carriers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Undergoing genetic testing at UVA for a personal or family history of breast or gynecologic cancers in Cancer Genetics.

Exclusion Criteria:

* Not receiving treatment at UVA
* Not English literate
* Unable to provide consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient population will be pulled from Gynecologic Oncology Women's Clinic and High Risk Breast and Ovarian Cancer Clinic at UVA
Enrollment: 20 (Estimated)
Dates: Start 2020-12-18 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Utility: Determine percentage of patients that report "GIA", the Genetic Information Assistant chatbox, is an acceptable form of family disclosure | 1 year
  Participants will complete a survey regarding the acceptability of GIA for use in disclosing results to family members. Feasibility will be assessed by tracking the number of family members contacted through GIA, the number of family members who access/interact with GIA, and the content topics most frequently covered in family member conversations.

SECONDARY OUTCOMES:
Impact:To determine percentage of family members that use the GIA chatbox by assessing the number of times GIA was used | 1 year
  Participants will complete a survey regarding the acceptability of GIA for use in disclosing results to family members. Feasibility will be assessed by tracking the number of family members contacted through GIA, the number of family members who access/interact with GIA, and the content topics most frequently covered in family member conversations.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ring KL, Bruegl AS, Allen BA, Elkin EP, Singh N, Hartman AR, Daniels MS, Broaddus RR. Germline multi-gene hereditary cancer panel testing in an unselected endometrial cancer cohort. Mod Pathol. 2016 Nov;29(11):1381-1389. doi: 10.1038/modpathol.2016.135. Epub 2016 Jul 22. PMID 27443514
- [Result] Walsh T, Casadei S, Lee MK, Pennil CC, Nord AS, Thornton AM, Roeb W, Agnew KJ, Stray SM, Wickramanayake A, Norquist B, Pennington KP, Garcia RL, King MC, Swisher EM. Mutations in 12 genes for inherited ovarian, fallopian tube, and peritoneal carcinoma identified by massively parallel sequencing. Proc Natl Acad Sci U S A. 2011 Nov 1;108(44):18032-7. doi: 10.1073/pnas.1115052108. Epub 2011 Oct 17. PMID 22006311
- See also: SGO Clinical Practice Statement: Screening for Lynch Syndrome in Endometrial Cancer — http://www.sgo.org/clinical-practice/guidelines/screening-for-lynch-syndrome-in-endometrial-cancer/
- See also: SGO Clinical Practice Statement: Genetic Testing for Ovarian Cancer — http://www.sgo.org/clinical-practice/guidelines/genetic-testing-for-ovarian-cancer/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/33/NCT04142333/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/33/NCT04142333/ICF_001.pdf